CLINICAL TRIAL: NCT02427152
Title: Pre-meal Planning and Expected Satiety
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Satt
Record Dates: First submitted 2015-03-18; First posted 2015-04-27 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Lean: body mass index: 18-25 kg/m²
- Overweight/Obese: body mass index: >25 kg/m²

SUMMARY:
Obesity is considered to be caused by an imbalance between energy expenditure and energy intake. A major determinant of our daily energy intake is the size of the meals that we consume. It has been suggested that decisions about portion sizes are often made in advance, before a meal begins. This pre-meal planning is considered to especially depend on the estimated 'expected satiety' and 'expected satiation' of different foods. Further, also factors like weight concern and palatability of the food might have their influence on meal size selection. In general, it is not clear how these factors are integrated during pre-meal planning and which brain networks are involved in these decisions/this process. Thus, the investigators plan to study pre-meal planning in healthy, normal-weight and overweight/obese individuals with functional magnetic resonance imaging under different cognitive instructions including pleasure, expected satiety and self-control in terms of health consequences. The investigators will explore the neural networks involved in pre-meal planning and expect them to be modulated by the before mentioned factors. Further, the investigators plan to explore gender differences and expect that female subjects will select smaller portion sizes especially in the self-control condition as they are often more concerned about their weight/health. Finally, the investigators will explore differences between lean and overweight subjects to elucidate factors that might lead to increased meal sizes in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* body mass index: 18-25 kg/m²; 25-35 kg/m²,
* right-handed,
* age: 18-35 years.

Exclusion Criteria:

* functional magnetic resonance imaging contraindications,
* claustrophobia,
* self-reported eating disorders,
* vegan or vegetarian diet, food allergies,
* intake of antidepressants,
* metabolic disorders.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: lean and overweight/obese healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Differential brain functions in reward, decision making and inhibitory control networks (brain functions will be measured by blood oxygen level dependent effects) | day 0
  brain functions will be measured by blood oxygen level dependent effects

SECONDARY OUTCOMES:
Differential behavioral measures of portion size selection | day 0

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, fMEG Center, Tübingen, Germany